

# Protocol number: **DS107G-02**

A RANDOMISED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PHASE II STUDY TO ASSESS THE EFFICACY AND SAFETY OF ORALLY ADMINISTERED DS107G TO PATIENTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS

Statistical Analysis Plan

**FINAL** 

Prepared by Josée Morin

Effective date: 19 OCT 2015

Version 1.0

# **SIGNATURE PAGE**

| Prepared by: | | |
|---|---|---|
| Josée Morin<br>Senior Biostatistician<br>Excelsus Statistics | Date | Signature |
| Approved by: | | |
| Annie Lévesque<br>Director, Scientific Affairs<br>Innovaderm Research Inc. | Date | Signature |
| Approved by: | | |
| Blánaid Ní Chuinneagáin<br>Clinical Scientist<br>Dignity Sciences | Date | Signature |

# **TABLE OF CONTENTS**

| SIC | SNATU | RE PAGE2 |
|-----|--------|-----------------------------------------------------------|
| TΑ | BLE O | F CONTENTS3 |
| LIS | T OF A | ABBREVIATIONS5 |
| 1 | Introd | duction |
| 2 | Study | Objectives7 |
| 3 | Study | / Methods7 |
| | 3.1 | General Study Design and Plan |
| | 3.2 | Inclusion-Exclusion Criteria and General Study Population |
| | 3.2.1 | Inclusion Criteria10 |
| | 3.2.2 | Exclusion Criteria1 |
| | 3.3 | Randomization and Blinding12 |
| | 3.4 | Study Variables12 |
| | 3.4.1 | Demographics and Baseline Characteristics12 |
| | 3.4.2 | Efficacy Variables13 |
| | 3.4.3 | Safety Variables18 |
| 4 | Samp | ole Size20 |
| 5 | Gene | eral Considerations |
| | 5.1 | Timing of Analyses |
| | 5.2 | Analysis Populations |
| | 5.2.1 | Intent-to-treat Population20 |
| | 5.2.2 | Safety Population20 |
| | 5.2.3 | Per-Protocol Population2 |
| | 5.3 | Missing Data/Multiple Observations |

| | 5.4 | Multi-centre Studies | 21 |
|----|--------|------------------------------------|----|
| | 5.5 | Multiple Testing | 22 |
| 6 | Sumr | mary of Study Data22 | 2 |
| | 6.1 | Subject Disposition | 22 |
| | 6.2 | Protocol Deviations | 23 |
| | 6.3 | Demographic and Baseline Variables | 23 |
| | 6.4 | Medical History | 23 |
| | 6.5 | Prior and Concomitant Medications | 23 |
| | 6.6 | Exposure and Treatment Compliance | 23 |
| 7 | Effica | ncy Analyses24 | 1 |
| | 7.1 | Primary Efficacy Analysis | 24 |
| | 7.2 | Secondary Efficacy Analyses | 24 |
| | 7.3 | Exploratory Efficacy Analyses | 25 |
| 8 | Safet | y Analyses25 | 5 |
| 9 | Repo | rting Conventions27 | 7 |
| 10 | Ted | chnical Details27 | 7 |
| 11 | Sui | mmary of Changes to the Protocol27 | 7 |
| 12 | Re | ferences27 | 7 |
| 13 | Мо | ck Tables, Listings and Figures28 | 3 |
| | 13.1 | Mock Tables | 28 |
| | 13.2 | Mock Listings | 66 |
| | 13 3 | Mock Figures | 99 |

### LIST OF ABBREVIATIONS

AD Atopic Dermatitis

AE Adverse Event/Adverse Experience

ANCOVA Analysis of Covariance

BMI Body Mass Index
BSA Body Surface Area
CI Confidence Interval
CRF Case Report Form
CS Clinically Significant

DGLA Dihomo-gamma-linolenic acid
DLQI Dermatology Life Quality Index
EASI Eczema Area and Severity Index

ICF Informed Consent Form

IGE Investigator's Global Evaluation of Eczema

ITT Intent-to-treat

IVRS Interactive Voice Response System
IWRS Interactive Web Response System
LOCF Last Observation Carried Forward

LLN Lower Limit of Normal

LLT Lower Level Term

MedDRA © Medical Dictionary for Regulatory Activities

NCS Non-clinically significant

POEM Patient Oriented Eczema Measure

PP Per Protocol

PT Preferred Term

SAE Serious Adverse Event/Serious Adverse Experience

SAF Safety Population

SAP Statistical analysis plan

SCORAD SCORing of Atopic Dermatitis

SD Standard Deviation

SOC System Organ Classification

TEAE Treatment-Emergent Adverse Event/Adverse Experience

TEWL Trans Epithelial Water Loss

ULN Upper Limit of Normal

WHODD World Health Organisation Drug Dictionnary

VAS Visual Analog Scale

### 1 Introduction

All statistical analyses will be performed in accordance with the protocol DS107G-02, dated 22-JUL-2015 (Version 2.2). This statistical analysis plan (SAP) includes a comprehensive and detailed description of the statistical methods and presentation of the data analysis by adding more details to the proposed methods in the protocol. The purpose of the SAP is to define the statistical approaches for the analysis of study data prior to database lock.

# 2 Study Objectives

<u>Primary objectives</u>: To compare the efficacy of orally administered DS107G capsules versus placebo, in the treatment of adult patients with moderate to severe atopic dermatitis.

<u>Secondary objective</u>: To assess the safety of orally administered DS107G capsules versus placebo, in adult patients with moderate to severe atopic dermatitis.

# 3 Study Methods

# 3.1 General Study Design and Plan

Approximately 100 patients with moderate to severe atopic dermatitis will be included in this multicenter, double-blind, placebo controlled, phase IIa study. All subjects will sign an informed consent and undergo screening for study eligibility. Subjects will be randomized (1:1) at baseline visit to either receive oral DS107G 2 g, or placebo once daily for 8 weeks in a fasting state.

Subjects will come to the clinic on 6 occasions: at screening, baseline, week 2, week 4, week 8 (end of treatment/early termination) and week 10 (follow-up). All subjects will exit the study at the Week 10 visit. The primary efficacy variable will be the proportion of patients achieving an IGA of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA at week 8. Secondary efficacy variables will include IGA at other visits, pruritus (obtained from the SCORAD visual analog scale), EASI, BSA, POEM, DLQI, SCORAD and TEWL (for selected sites only). Safety will be assessed through adverse events, physical examination, vital signs and safety laboratory tests (including pregnancy tests for women of childbearing potential). Pharmacokinetic samples will be obtained at Baseline (Day 0), week 4 and week 8 visits in order to measure total and free DGLA plasma trough levels. A separate plasma sample will be retained for later analysis of total fatty acid profile and interleukin profile.

The study flow chart of all assessment and timing is presented in Figure 1.

Figure 1. Study Flow Chart

| Visit | Screening | Baseline | Week 2 | Week 4 | Week 8 /<br>ET visit | Follow up<br>visit / Week<br>10 |
|---|---|---|---|---|---|---|
| Day | -30 to -1 | 0 | 14 (± 2) | 28 (± 2) | 56 (± 2) | 70 (±3) |
| Informed Consent | Х | | | | | |
| Demographics | Х | | | | | |
| Medical / Surgical History | Х | Х | | | | |
| Ongoing medical history <sup>y</sup> | | | | | Х | Х |
| Review Inclusion/Exclusion Criteria | Х | Х | | | | |
| Hanifin and Rajka criteria | Х | | | | | |
| Assign subject identifier number | Х | | | | | |
| Randomization | | Х | | | | |
| Concomitant Medications | Х | Х | Х | Х | Х | Xδ |
| Safety labs and inflammation<br>biomarkers: Serum Chemistry<br>(including FSH levels at screening<br>when applicable* and interleukin<br>profile), Coagulation, Hematology,<br>urinalysis | ΧΦ | x | | x | x | <b>(X**)</b> <sup>Φ, δ</sup> |
| Pharmacokinetics (pre-dose blood draw) <sup>††</sup> | | Х | | х | х | |
| Blood draw for fatty acid profile sample <sup>††,</sup> | | Х | | х | X | |
| Pregnancy Test (β-hCG if female of childbearing potential)* | x | X | х | х | X | Xδ |
| Vital Signs | X | X | X | X | Х | Xδ |
| Physical Examination | X | | | X | X | <b>X</b> 8 |
| ВМІ | X | X | | | X | |
| Study Drug Administration (on site) <sup>€</sup> | | X | | X | § | |
| Dispense Study Drug | | Х | Х | Х | | |
| Collect Study Drug | | | X | X | X | |
| Dispense Subject Compliance Log | | X | X | X | | |
| Collect and Review Subject<br>Compliance Log | | | х | X | X | |
| Capsule count | | | X | X | X | |
| BSA | X | X | X | X | X | X |
| IGA | Х | Х | Х | Х | Х | Χ |
| EASI assessment | | X | Х | Х | Х | X |
| SCORAD assessment / VAS pruritus assessment | | Х | х | х | х | x |
| POEM questionnaire | | Х | Х | Х | Х | Х |
| DLQI questionnaire | | Х | Х | Х | Х | Х |
| TEWL (selected sites only) | | Х | Х | Х | Х | Х |
| Adverse Events† | | X <sup>†</sup> | Х | Х | Х | Xδ |

<sup>¥::</sup> For women greater than 40 and less than 60 years of age who have had a cessation of menses for at least 12 months but less than 24 months

<sup>\*\*:</sup> Only if clinically significant change from baseline in safety lab results at week 8

- \*: Serum pregnancy test at screening and week 8 / ET visits, urine test pregnancy for all other visits
- ††: If a subject took study medication prior to the visit, he/she will be required to come back the following day for PK blood draws.
- €: Subjects must be fasting for at least 8 hours before and 60 minutes after drug administration
- §: Subjects will be instructed to take their last study drug dose the day preceding week 8 visit.
- †: Collection of AE will start after the first study drug administration
- Y: Assessment if any ongoing condition has improved since baseline.
- Φ: Interleukin profile will not be evaluated at screening and week 10.
- $\delta$ : In the case the subject ends the study before completion, the subject will also return 2 weeks after the ET visit for safety assessment listed at Week 10.

### 3.2 Inclusion-Exclusion Criteria and General Study Population

To participate in the study, subjects must meet all the inclusion criteria and none of the exclusion criteria.

#### 3.2.1 Inclusion Criteria

Subjects must meet all of the following criteria to be eligible for this study:

- Male or female subject aged 18 years and older on the day of signing the informed consent form (ICF).
- Clinically confirmed diagnosis of active atopic dermatitis according to Hanifin and Rajka criteria.
- Moderate to severe atopic dermatitis at baseline as defined by an IGA of minimum 3 at baseline visit.
- Atopic dermatitis covering minimum 10% of the body surface area at baseline.
- Body mass index (BMI) is between 18 and 35 kg/m<sup>2</sup> inclusively.
- Female patients of childbearing potential must use adequate contraception or have a sterilized partner for the duration of the study: systemic hormonal contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicide, or agree to sexual abstinence. Hormonal contraceptives must be on a stable dose for at least one month before baseline. Note: Women of non-child bearing potential are:
  - women who have had surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation)
  - women greater than 60 years of age
  - women greater than 40 and less than 60 years of age who have had a
    cessation of menses for at least 12 months and a follicle-stimulating hormone
    (FSH) test confirming non-childbearing potential (FSH ≥40 mIU/mL) or
    cessation of menses for at least 24 months without FSH levels confirmed.
- Patients who are able and willing to stop treatment for atopic dermatitis throughout the study (except for allowed emollients).
- Capable and willing to give signed informed consent and the consent must be obtained prior to any study related procedures.

#### 3.2.2 Exclusion Criteria

Subjects must not have the following to be eligible for this study:

- Female patients with positive pregnancy test at screening or Day 0 visit (baseline) or lactating women.
- Any clinically significant controlled or uncontrolled medical condition or laboratory abnormality that would, in the opinion of the investigator, put the patient at undue risk or interfere with interpretation of study results.
- Clinically significant impairment of renal or hepatic function.
- Other skin conditions that might interfere with atopic dermatitis diagnosis and/or evaluation (such as psoriasis or current viral, bacterial and fungal skin infections).
- History of hypersensitivity to any substance in DS107G or placebo capsules.
- Use of biologics 3 months prior to start of treatment/ Day 0 visit (baseline), or 5 half-lives (whichever is longer).
- Use of systemic treatments (other than biologics) that could affect atopic dermatitis
  less than 4 weeks prior to baseline visit (Day 0), e.g. retinoids, calcineurin inhibitors,
  methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and
  oral/injectable corticosteroids; Intranasal corticosteroids and inhaled corticosteroids
  for stable medical conditions are allowed.
- Treatment with any experimental drug within 30 days prior to Day 0 visit (baseline), or 5 half lives (whichever is longer).
- Excessive sun exposure, use of tanning booths or other ultraviolet (UV) light sources
   4 weeks prior to Day 0 visit (baseline) and/or is planning a trip to sunny climate to use tanning booths or other UV sources between screening and follow-up visits.
- Use of any topical medicated treatment for atopic dermatitis 2 weeks prior to start of treatment/Day 0 visit (baseline), including but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials and bleach baths.
- Use of topical products containing urea, ceramides or hyaluronic acid for 2 weeks prior to Day 0.
- Use of anti-histamines for atopic dermatitis within 2 weeks of baseline.
- Significant uncontrolled cardiovascular (a history of ECG abnormalities that are clinically significant in the opinion of the investigator), neurologic, malignant, psychiatric, respiratory or hypertensive disease, as well as diabetes and arthritis.
- Medical history of chronic infectious disease (e.g., hepatitis B, hepatitis C or infection with human immunodeficiency virus).
- History of clinically significant drug or alcohol abuse in the last year prior to Day 0 (baseline).

# 3.3 Randomization and Blinding

Approximately 100 patients will be randomized into double-blind treatment groups a 1:1 ratio by an Interactive Web Response System (IWRS) or Interactive Voice Response System (IVRS), as follows:

- Treatment group A: 2 grams DS107G (4 capsules)
- Treatment group B: 2 grams placebo capsules (4 capsules)

A randomization list permuted blocks will be generated by Dignity Sciences or its designee. The randomization schedule with study drug assignments will be generated prior to the start of the study and will be known only to the individuals responsible for labeling the study drug. The IVRS or IWRS will assign a study drug kit number to each subject and the contents will be based on the randomization code.

Each subject will be assigned a patient identifier number during screening that will be used on all patient documentation. The patient identifier number will contain the site number and the patient number assigned in numerical order at the screening visit (e.g.: 02-010 for the tenth patient screened at the site #02). Numbers will be assigned in ascending order starting with 001.

Four patients were randomized under site 6X instead of site 06 (6X-001, 6X-002, 6X-004 and 6X-005). Those 4 patients will be reassigned to site 06 for the presentation and the summarization of the results.

# 3.4 Study Variables

### 3.4.1 Demographics and Baseline Characteristics

**Age** calculated in years is defined as the difference between the informed consent date and the birthdate.

**Gender** is a code list where 1 equals Male and 2 equals Female.

**Height** in centimeters measured to the nearest centimeter.

**Weight** in kilograms (kg) measured to one decimal place.

**Body Mass Index (BMI)** will be calculated as the weight (kg) divided by the square of height (m) and rounded to one decimal place (kg/m<sup>2</sup>).

**Race** is an integer ranging from 1 to 6, where 1 corresponds to American Indian or Alaska Native, 2 corresponds to Asian, 3 corresponds to Black or African American, 4 corresponds to Native Hawaiian or Other Pacific Islander, 5 corresponds to White, and 6 corresponds to Other.

**Ethnicity** is code list where 1 corresponds to 'Hispanic or Latino' and 2 corresponds to 'Not Hispanic or Latino'.

#### **Medical History**

Medical history will be coded using the Body System Code as the following: Eyes-Ears-Nose-Throat, Respiratory (Asthma/Other), Cardiovascular, Gastrointestinal, Hepatobiliary, Genitourinary/ Renal, Reproductive, Neurological, Endocrine, Hematological, Musculoskeletal, Dermatologic, Extremities, Immunological, Psychiatric, and Allergies.

#### Medications

Medications will be coded using the Preferred Term from the WHO Drug Dictionary (Sept-2014 B2). If the start and end dates of the medication are prior to the study drug start date then the medication will be coded as prior medication. Otherwise the medication will be considered as concomitant medications.

### 3.4.2 Efficacy Variables

### 3.4.2.1 Primary Efficacy Variable

The primary efficacy variable is the **Investigator's Global Assessment (IGA)** of Disease Severity and will be assessed at each visit. The IGA is a global assessment of the current state of the disease. It is a 6-point morphological assessment of overall disease severity and will be determined according to the following definitions:

| Score | Grade | Definition |
|---|---|---|
| 0 | Clear | No evidence of disease with the exception of residual pigment changes and/or xerosis |
| 1 | Almost clear | Perceptible erythema, papulation/infiltration |
| 2 | Mild | Mild erythema, papulation/infiltration |
| 3 | Moderate | Moderate erythema, papulation/infiltration |
| 4 | Severe | Severe erythema, papulation/infiltration |
| 5 | Very Severe | Severe erythema, papulation/infiltration with oozing/crusting |

Change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.

The IGA will be also examined using the following criteria:

- IGA of 0 (clear) or 1 (almost clear) at Week 8;
- at least a 2-point decrease in IGA at Week 8;
- at least a 1-point decrease in IGA at Week 8;
- No Change or Increased from Baseline in IGA at Week 8

#### 3.4.2.2 Secondary Efficacy Variable

Secondary efficacy variables are as follows:

 The Eczema Area and Severity Index (EASI) will be assessed at each visit, except screening visit. It quantifies the severity of a subject's atopic dermatitis based on both lesion severity and the percent of BSA affected.

Four anatomic sites – head, upper extremities, trunk, and lower extremities – are assessed for erythema, induration (papules), excoriation and lichenification as seen on the day of the examination. The severity of each sign is assessed using a 4-point scale: 0 = No symptoms, 1 = Slight, 2 = Moderate, 3 = Marked.

The area affected by atopic dermatitis within a given anatomic site is estimated as a percentage of the total area of that anatomic site and assigned a numerical value according to the degree of atopic dermatitis involvement as follows: 0 = no involvement, 1 = < 10 %, 2 = 10 to < 30%, 3 = 30 to < 50%, 4 = 50 to < 70%, 5 = 70 to < 90%, 6 = 90 to 100 %.

The EASI score is obtained by using the formula:

EASI = 
$$0.1 * (E_h + I_h + Ex_h + L_h) * A_h +$$
  
 $0.2 * (E_u + I_u + Ex_u + Ex_u) * A_u +$   
 $0.3 * (E_t + I_t + Ex_t + Ex_t) * A_t +$   
 $0.4 * (E_l + I_l + Ex_l + Ex_l) * A_l$ 

Where E, I, Ex, L and A denote erythema, induration, excoriation, lichenification and area, respectively, and h, u, t, and I denote head, upper extremities, trunk, and lower extremities, respectively. The EASI score ranges from 0 (no disease) - 72 (maximal disease). The score will be set to missing in case of at least one missing value.

The change from baseline in EASI at Week 2, Week 4, Week 8, and Week 10 will be calculated as the value at the visit minus the value at Baseline. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.

• The overall Body Surface Area (BSA) affected by AD will be evaluated (from 0 to 100%) at each visit. One patient's palm represents 1% of his/her total BSA. For all study visits except at screening, the BSA of involved skin will be measured with the SCORAD measurement. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8 and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.

• The SCORing Atopic Dermatitis (SCORAD) will be measured at each visit, except the screening visit. The SCORAD grading system is a standard tool to assess the AD severity in clinical studies in Europe. Six items (erythema, edema/papulation, oozing/crusts, excoriation, lichenification, and dryness) are selected to evaluate the AD severity. The intensity of each item is graded using a 4-point scale: 0 = No symptoms, 1 = Mild, 2 = Moderate, 3 = Severe.

The area chosen for grading must be representative (average intensity) for each item. The individual intensity ratings for each item will then be added (ranging from 0-18) and multiplied by 3.5, giving a maximal score of 63.

The overall BSA affected by AD is evaluated (from 0 to 100%) and divided by 5. One patient's palm represents 1% of his/her total BSA. The maximum is 20.

Subjective items include loss of sleep and the occurrence of pruritus. These are evaluated by asking patients to indicate on the 10-cm scale (0-10) of the assessment form the point corresponding to the average value for the last three days/nights. The combined maximum score of these two is 20.

The sum of the above measures represents the SCORAD which can vary from 0 to 103. If the subjective scores of pruritus and loss of sleep are excluded, the SCORAD becomes objective SCORAD (score range 0-83).

The score will be set to missing if there is at least one missing value. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.

- The Visual Analog Scale (VAS) of Pruritus will be assessed with the SCORAD measurement for all study visits except screening. This will be evaluated by asking subjects to indicate on the 10-cm scale (0-10) of the assessment form the point corresponding to the average value for the last three days/nights. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.
- The **Patient-Oriented Eczema Measure (POEM)** will be assessed at each visit, except screening visit. The POEM is a self assessment of disease severity by the patient. The following questions are to be rated as: 0=No Days, 1=1-2 Days, 2=3-4 Days, 3=5-6 Days, 4=Everyday.

- 1. Over the last week, on how many days has your skin been itchy because of your eczema?
- 2. Over the last week, on how many nights has your sleep been disturbed because of your eczema?
- 3. Over the last week, on how many days has your skin been bleeding because of your eczema?
- 4. Over the last week, on how many days has your skin been weeping or oozing clear fluid because of your eczema?
- 5. Over the last week, on how many days has your skin been cracked because of your eczema?
- 6. Over the last week, on how many days has your skin been flaking off because of your eczema?
- 7. Over the last week, on how many days has your skin felt dry or rough because of your eczema?

The POEM score is the sum of the 7 question ratings for a possible total of 28 (more severe eczema). The score will be set to missing if there is at least one missing value. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated

 The Dermatology Life Quality Index (DLQI) questionnaire is a simple 10-question validated questionnaire which will be completed at each visit, except screening. The following questions are to be assessed by the patient:

| 1. | Over the last week, how itchy, sore, painful or | Very much (3) | |
|---|---|---|---|
| | stinging has your skin been? | A lot (2) | |
| | gang nac year came com | A little (1) | |
| | | Not at all (0) | |
| 2. | Over the last week, how embarrassed or self | Very much (3) | |
| | conscious have you been because of your skin? | A lot (2) | |
| | | A little (1) | |
| | | Not at all (0) | |
| 3. | Over the last week, how much has your skin | Very much (3) | |
| | interfered with you going <b>shopping</b> or looking | A lot (2) | |
| | after your home or yard? | A little (1) | |
| | | Not at all | Not relevant (0) |
| 4. | Over the last week, how much has your skin | Very much (3) | |
| | influenced the <b>clothes</b> you wear? | A lot (2) | |
| | | A little (1) | |

| | | Not at all | Not relevant (0) |
|---|---|---|---|
| 5. | Over the last week, how much has your skin affected any <b>social</b> or <b>leisure</b> activities? | Very much (3)<br>A lot (2)<br>A little (1)<br>Not at all | Not relevant (0) |
| 6. | Over the last week, how much has your skin made it difficult for you to do any <b>sport</b> ? | Very much (3)<br>A lot (2)<br>A little (1)<br>Not at all | Not relevant (0) |
| 7. | Over the last week, has your skin prevented you from <b>working</b> or <b>studying</b> ? | Yes (3)<br>No (0) | |
| | If "No", over the last week how much has your skin been a problem at <b>work</b> or <b>studying</b> ? | A lot (2)<br>A little (1)<br>Not at all (0) | |
| 8. | Over the last week, how much has your skin created problems with your <b>partner</b> or any of your <b>close friends</b> or <b>relatives</b> ? | Very much (3)<br>A lot (2)<br>A little (1)<br>Not at all | Not relevant (0) |
| 9. | Over the last week, how much has your skin caused any <b>sexual difficulties</b> ? | Very much (3)<br>A lot (2)<br>A little (1)<br>Not at all | Not relevant (0) |
| 10 | Over the last week, how much of a problem has the <b>treatment</b> for your skin been, for example by making your home messy, or by taking up time? | Very much (3)<br>A lot (2)<br>A little (1)<br>Not at all | Not relevant (0) |

The DLQI score is the sum of the 10 questions for a possible total of 30 (quality of life is impaired). 'Not relevant" and "Unanswered' questions will be scored as 0. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated

 Trans epidemal Water Loss (TEWL), the clinical severity of AD and associated effect on skin barrier function will be evaluated at each visit, except the screening visit. This evaluation will be performed at selected sites that have demonstrated previous experience with this device.

At Baseline (Day 0), the investigator will select three representative areas of active AD for each subject; the location of these sites will be recorded. At subsequent visits, TEWL readings for each area of AD will be taken in standard room ambient conditions (22-25°C, 40-60% relative humidity); the mean of the TEWL measurements will be used for the

analyses. The change from Baseline will be calculated as the value at the visit minus the value at Baseline. The change from baseline will be calculated at Week 2, Week 4, Week 8, and Week 10. Percent change from baseline will also be calculated. In addition, change and percent change from Week 8 to Week 10 will be calculated.

### 3.4.3 Safety Variables

#### 3.4.3.1 Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as AEs that developed, worsened or became serious after the first dose of study drug during the study, i.e. from the study drug start date to the end of study.

TEAEs will be coded according to Medical Dictionary for Regulatory Activities (MedDRA, version 17.0) terminology. The coding process using MedDRA will be conducted by the data management where lower level term (LLT), the preferred term (PT) and system organ class (SOC) will be assigned to each AE term.

Descriptions of AEs will include the date of onset, the date the AE ended (if it resolved), the severity and seriousness of the AE, the relationship of the AE to study medication, and the outcome. If the onset date of the AE is incomplete or missing and the end date is incomplete or missing, or the end date is after the start of treatment, then the event will be evaluated as a TEAE. If the start date is at the Baseline Visit and the end date is incomplete or missing, then the event will be evaluated as a TEAE. The AE onset will also be shown relative (in number of days) to the day of first dose.

### 3.4.3.2 Laboratory Safety Variables

Urinalysis, hematology (with differential and coagulation testing), a standard chemistry panel (chemistry includes liver function tests and cholesterol), coagulation, and serum pregnancy test for women of childbearing potential will be collected during the study (see Figure 1. Study Flow Chart for details). The list of laboratory parameters are presented in Table 1 below.

Table 1. Clinical laboratory Testing

| Laboratory testing | Tests included |
|---|---|
| Hematology | Basophils, Eosinophils, HCT, HGB, Lymphocytes, MCH, MCV, Monocytes, Neutrophils, platelets, RBC, WBC |
| Coagulation | APTT, INR, PT |
| Serum Chemistry | Albumin, Alkaline Phosphatase, ALT, AST, Chloride, Cholesterol (non-fasting), CK, Creatinine (Enzymatic), GGT, Glucose Random, LDH, Potassium, Sodium, Total Bilirubin, Triglycerides, Urea (BUN), Uric Acid β-hCG for females of childbearing potential |
| Urinalysis | Blood, Glucose, pH, Protein |

Laboratory results will be transferred by the laboratory itself. The data will include the visit date and time, the laboratory result type (e.g. hematology), the analyte name, the result, the unit, the reference values, and the abnormal flag.

#### 3.4.3.3 Vital Signs

Vital signs will be assessed at each visit and include systolic and diastolic blood pressure, pulse, oral temperature and respiratory rate. The following variables were created for each vital sign.

- Value at the time specified is the value specified for the parameter on the CRF
- Change from baseline is the value at the time specified minus the value at baseline

#### 3.4.3.4 Physical Examination

The following sites/systems will be included in the Physical examination. Each system will be scored as: Normal, Abnormal Not Clinically Significant, or abnormal clinically significant.

- General appearance
- Dermatological (except atopic dermatitis)
- Head, Eyes, Ears, Nose, Throat (HEENT)

- Respiratory
- Cardiovascular
- Abdominal
- Neurological
- Musculoskeletal
- Lymphatic

### 3.4.3.5 Total and Free DGLA plasma levels, Total Fatty Profile and Interleukins levels

Total DGLA and free DGLA trough plasma levels will be measured at Baseline, week 4 and week 8. Total fatty profiles and interleukins levels will not be covered in this SAP.

### 4 Sample Size

The primary endpoint can be translated as a responder analysis where a subject will be classified as Responder if he/she achieves an IGA score of 0 (clear) or 1 (almost clear) at Week 8, considering a 2-point decrease from baseline. A sample size of 45 subjects will have a power of 80% to detect a statistically significant difference of 25% between responders from treated group and from the placebo group, based on a chi-square test and an alpha of 0.05. Based on the literature review, it is expected that the placebo could reach up to 7%, so the minimal proportion expected in the treated group should be at least 32%. Allowing for 10% drop-out, a total of 100 subjects should be enrolled in the study.

### 5 General Considerations

# **5.1 Timing of Analyses**

The final analysis will be performed on data transferred to the statistician, having been documented as meeting the cleaning and approval requirements of the database lock and after the finalisation and approval of this SAP document.

There is no interim analysis planned for this study.

# 5.2 Analysis Populations

#### 5.2.1 Intent-to-treat Population

The Intent-to-treat (ITT) population will consist of all randomized subjects. Analysis will be done according to the randomized treatment. This population will be used for all efficacy analyses.

#### 5.2.2 Safety Population

The safety population will be defined as all randomized subjects who received at least one dose of the medication. Analysis will be done according to the actual treatment subjects received.

#### 5.2.3 Per-Protocol Population

The per-protocol (PP) population will include all subjects who received at least one dose of the medication and who had at least one post-baseline evaluation on the primary endpoint of IGA with no significant protocol deviations. Analysis will be done according to the actual treatment subjects received.

Protocol deviation will be listed and summarized. Prior to database lock, significant protocol deviation will be defined and reviewed in a blinded fashion conjointly by the medical director (or delegate) and the statistician. Patients with significant protocol deviations will be excluded from the PP population.

The PP population will be used for all efficacy analyses as supportive analyses.

### 5.3 Missing Data/Multiple Observations

No imputation will be done for all population and all parameters, except for the primary endpoint. A supportive analysis using the last observation carried forward (LOCF) method will be performed on responder analysis (see section 7.1 for details).

In the event that two values were collected for the same visit, the scheduled assessment value will be retained in the analyses, unless otherwise specified (e.g. lab error). However, all values will be presented in the data listings. Laboratory values of '< X' ou '> X' will be set to 'X' for the analysis.

### 5.4 Multi-centre Studies

The primary efficacy analysis will be performed with site included in the statistical model as a stratification factor. A sensitivity analysis will also be conducted without site. Analysis on the secondary efficacy endpoints will include information on site. Safety data will be presented with all study sites pooled. Safety analysis will be performed with data from all sites being pooled.

To obtain a sufficient and better-balanced number of subjects among study sites, pooling of study sites will be applied prior to performing the statistical inference and unblinding treatment. Sites without at least 5 subjects in the ITT population will be incorporated into pooled sites as follows:

- All such sites with less than 5 subjects will be ordered from the lowest to the highest in terms of number of ITT subjects. In case of ties, the ordering for tied sites will be determined according to the site identification number (from smallest to largest).
- Sites will be combined beginning at the smallest until the resulting pooled site contains at least 5 ITT subjects. The sites pooled in this way will be considered as a single site in the statistical analyses.
- The process described above will resume for the remaining sites not meeting the criterion of at least 5 subjects. If the final set of pooled site does not meet the criterion of at least 5 ITT subjects, the final set will be pooled with the preceding pooled site.

### 5.5 Multiple Testing

Since there are only 2 treatment groups involved in this study, no correction for multiplicity will be performed.

### 6 Summary of Study Data

All continuous variables will be summarised using the following descriptive statistics: n (non-missing sample size), mean, standard deviation (SD), median, inter-quartile range (25th and 75th percentiles), maximum, and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures.

In general, all data will be listed, sorted by treatment group, site and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for each treatment in the same order (DS107G, Placebo) and will be annotated with the total population size relevant to that table/treatment.

Day 0 is the first day of study medication. In the event that there is more than one value for a given assessment prior to the study drug start date, the value obtained closest to Day 0, before administration of study drug will be considered as the baseline value. The baseline value will be the value nearest to and before the first dose of the study medication.

All statistical tests will be two-sided and will be performed with a significant level of 0.05, unless otherwise specified.

# **6.1 Subject Disposition**

Subject disposition information, including the counts and percentages of subjects screened, screen failed, randomized, and who completed the study will be summarized based on all enrolled subjects (i.e. who signed the informed consent form).

Tables will be created indicating the number of subjects by treatment group in each of the analysis populations and attending each visit. Finally, for each of the analysis populations there will be tables indicating by treatment group the number of days in the study, the percentage of subjects discontinued and the reasons for discontinuation. Overall comparability of subject's discontinuation between the two treatment groups will be tested using a Fisher exact test and overall comparability of the reasons for discontinuation for both treatment groups will be done using an exact Pearson's Chi-Squares test.

Number of days in the study will be calculated as the difference between the date of the last visit (Follow up/Week 10) and the informed consent date plus 1.

### 6.2 Protocol Deviations

Protocol deviations may include, but are not limited to:

- Visit outside of the visit window
- Missed visit
- Missed/Extra dose(s)
- Study Procedure(s) not done
- Prohibited medication
- Etc.

A listing of all protocol deviations will be presented and documented in the study file. A descriptive summary table of protocol deviation categories by treatment group will be presented.

### 6.3 Demographic and Baseline Variables

Demographic and baseline variables will be analysed using descriptive statistics.

### 6.4 Medical History

Medical history will be presented using the frequency and percentage of subject by Body System Code.

### 6.5 Prior and Concomitant Medications

Medications will be coded to the preferred generic name using the WHO-Drug dictionary (version June 2013 B2). Compound product will be coded to the brand name. Any medications that started and ended prior to the study drug start date will be considered as "Prior" and "Concomitant", otherwise. A listing of all medications will be produced.

# 6.6 Exposure and Treatment Compliance

Descriptive statistics will be presented by Treatment group on the extent of exposure and the compliance.

The extent of exposure will be defined as:

Number of days on drug = Date of Week 8/ET Visit – First dose study drug administration date.

Compliance will be calculated as follows:

$$\frac{\text{(Sum of all capsules dispensed)} - \text{(Sum of all capsules returned)}}{\text{(4} \times \text{Number of days on drug)}} * 100$$

# 7 Efficacy Analyses

All efficacy variables will be summarized using descriptive statistics by treatment group at each visit.

# 7.1 Primary Efficacy Analysis

The primary endpoint can be translated as a responder analysis where a subject will be classified as Responder if he/she achieves an IGA score of 0 (clear) or 1 (almost clear) at Week 8, considering a 2-point decrease from baseline. Patients who did not complete the study (i.e. subjects with an early termination visit at Week 8) will be classified as non-responder.

The comparison between groups for the primary endpoint will be done using a Cochran-Mantel–Haenszel (CMH) test where the site will be used as the stratification factor. A sensitivity analysis will also be conducted using a Fisher's exact without Site. Subgroup analyses will also be performed on responders vs. non responders (using CMH test stratified for site) for each subgroup of patients (Very Severe/Severe and Modreate), separately.

The primary efficacy analysis will be done using observed values. A supportive analysis will be conducted using the LOCF method. For subjects who did not complete the study, the last non-missing IGA results (including results collected during the early termination Week 8 visit) will be used.

The analyses will be done using the ITT population and will serve as the primary analysis while the analysis of the primary endpoint using the PP population will be used as a supportive analysis.

# 7.2 Secondary Efficacy Analyses

The second efficacy endpoints are:

- Change from baseline in IGA at week 2, 4, and 8
- Change from baseline in EASI at week 2, 4, and 8
- Change from baseline in POEM at week 2, 4, and 8
- Change from baseline in DLQI at week 2, 4, and 8
- Change from baseline in SCORAD at week 2, 4, and 8
- Change from baseline in VAS at week 2, 4, and 8
- Change from baseline in BSA at week 2, 4, and 8
- Proportion of patients achieving at least 1-point decrease in IGA at Week 8

All secondary endpoint based on the change from baseline will be assesd using an ANCOVA where the change from baseline will be the dependant variable and including the treatment group and site as fixed effects and baseline value as a covariate. In addition, ANCOVA will also be performed on the change from baseline at week 10 and on the change from Week 8 to Week 10.

All secondary endpoint based on categories will be analysed using a Cochran–Mantel–Haenszel test stratified by site and the p-value from this test will be presented along with frequency and percentage of subjects for each category.

All change and percent change values will be summarized using descriptive statisitics, for each treatment group and visit. Proportion of subjects with no, 1-point, 2-point, 3-point, decrease/increase, will be presented at Week 8.

All statistical analyses will de bone at each visit and using the ITT (primary analysis) and PP (supportive analysis) population. All the analyses will be done using observed values. Results collected during the early termination visit related to Week 8 and Week 10 will not be included. No sensitivity analysis will be done for missing values.

# 7.3 Exploratory Efficacy Analyses

Change from baseline in TEWL at week 2, 4, and 8 will be analyzed using an ANCOVA as described in section 7.2.

# 8 Safety Analyses

Safety analysis will be performed based on the safety analysis population. No inferential statistics will be done on safety variables.

### Adverse Events

Treatment-emergent AEs (TEAEs) will be summarized by the number of subjects reporting the events, as well as by System Organ Class, Preferred Term, severity, seriousness, and relationship to study medication. A general summary table will be provided with the number of TEAEs, Related TEAEs, Serious TEAEs and Serious Related TEAEs.

For the summary of TEAEs by severity, each patient will be counted only once within a System Organ Class or a Preferred Term by using the TEAEs with the highest intensity within each category for each analysis. For the summary of TEAEs by relationship to study medication, each patient will be counted only once within a System Organ Class or a Preferred Term by using the AEs with the greatest reported relationship within each category. For the summary of AEs by relationship to study medication and severity, each patient will be counted only once within a System Organ Class or a Preferred Term by using (1) the greatest reported relationship followed by (2) the highest reported intensity.

The following tables will be presented:

- TEAEs by SOC/PT;
- Related TEAEs by SOC/PT;
- TEAEs by severity and SOC/PT;
- TEAEs by relationship and SOC/PT;
- TEAEs by relationship/severity and by SOC/PT;
- TEAEs leading to treatment discontinuation by SOC/PT
- Serious TEAEs (SAEs) by SOC/PT;
- Related Serious TEAEs by SOC/PT;

### **Clinical Laboratory**

The clinical laboratory results (including value at visit and change from baseline) will be presented descriptively for each time point. Shift table from baseline to each post-dose time points will be presented.

### Vital Signs

The vital signs (including value at visit and change from baseline) will be presented descriptively for each time point.

### Total and Free DGLA plasma levels, Total Fatty Profile and Interleukins levels

Relationship between DGLA levels and the severity of disease will be looked at. A scatter plot of Total and Free DGLA concentrations at baseline versus IGA score at Week 8 and versus change from baseline in IGA at Week 8 will be produced by treatment group as well as for both treatment combined. Spearman correlation coefficient will be presented. In addition, change from Baseline in DGLA versus change from baseline in IGA will also be plotted (along with Spearman correlation coefficient) at Week 8 as well as the change from baseline in DGLA at Week 8 versus the change from baseline in IGA at Week 10.

Descriptive statistics of level of DGLA will be presented by treatment, visit and responder status.

The analysis of the total fatty and interleukins data will not be covered in this SAP.

# 9 Reporting Conventions

P-values will be reported to 3 decimal places. If value is less than 0.001, then it will be shown as "<0.001". The mean, SD, Median and inter-quantile will be reported to one decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data.

### 10 Technical Details

All statistical processing will be performed using SAS® software, Version 9.2, or higher.

# 11 Summary of Changes to the Protocol

Additional analyses (not included in the protocol) were added in the statistical analysis plan.

- Total and Free DGLA plasma level in relation with IGA results
- Respondeur analysis controlling for the information on IGA at Baseline
- Comparability of the discontinuation rates and of the reasons for discontinuation for both treatment groups

### 12 References

No applicable.

# 13 Mock Tables, Listings and Figures

All tables, listings and figures (TLF) will be generated through SAS.

The title will be unique for each TLF and self-explanatory. The header section will comprise of the Sponsor's name, the protocol number, the TLF number, the TLF title, the analysis population, and the page number (Page X of Y). The footer section of the table will include the date and time of the execution of the program, and the name of the program. All necessary footnotes will be provided to add clarity to the TLF.

The font will be "Courier New", 8-9 points, or similar. The orientation will be landscape with 1 inch margins. The tables and figures will be placed under Appendix 14 in the Clinical Study Report while the listings will be placed in the Appendix 16.

The following sections display the expected TLFs. All efforts were made to create representative mock TLFs, however, these may change depending on the format and layout of the data, without changing the purpose of the presentation. In the event a major change to a TLF is required, this will be discussed within the study team and necessary documentation will be created.

### 13.1 Mock Tables

The list of tables is presented in the table below followed by the actual mock tables.

| Table Number | Title | Population |
|---|---|---|
| | Study Conduct Tables | |
| 14.1.1 | Summary of Subject Enrollment and Disposition | All |
| 14.1.2 | Summary of Visits Completed | SAF/ITT/PP |
| 14.1.3 | Summary of Study Completion | SAF/ITT/PP |
| 14.1.4 | Summary of Protocol Deviations | SAF |
| 14.1.5.1/.2/.3 | Summary of Subject Demographics and Baseline Characteristics | SAF/ITT/PP |
| 14.1.6 | Summary of Medical History | SAF |
| 14.1.7.1/.2/.3 | Summary of Study Drug Exposure and Compliance | SAF/ITT/PP |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

| Table Number | Title | Population |
|---|---|---|
| | Efficacy Tables | |
| 14.2.1.1.1 | Summary of Investigator's Global Assessment – Responder Analysis at Week 8 | ITT |
| 14.2.1.1.2 | Summary of Investigator's Global Assessment – Responder Analysis at Week 8 | PP |
| 14.2.1.1.3 | Summary of Investigator's Global Assessment – Responder Analysis at Week 8 – Supportive Analysis (LOCF) | ITT |
| 14.2.1.1.4 | Summary of Investigator's Global Assessment – Responder Analysis at Week 8 - Supportive Analysis (LOCF) | PP |
| 14.2.1.2.1 | Summary of Investigator's Global Assessment – Actual, Change and Percent Change from Baseline | ITT |
| 14.2.1.2.2 | Summary of Investigator's Global Assessment – Actual, Change and Percent Change from Baseline | PP |
| 14.2.1.3.1 | Summary of Investigator's Global Assessment – Proportion of Subjects with at least 1-point decrease, and with no or increase/decrease at Week 8 | ITT |
| 14.2.1.3.2 | Summary of Investigator's Global Assessment – Proportion of Subjects with at least 1-point decrease, and with no or increase/decrease at Week 8 | PP |
| 14.2.2.1 | Summary of Eczema Area and Severity Index – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.2.2 | Summary of Eczema Area and Severity Index – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.3.1 | Summary of Patient-Oriented Eczema Measure – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.3.2 | Summary of Patient-Oriented Eczema Measure – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.4.1 | Summary of Dermatology Quality of Life Index – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.4.2 | Summary of Dermatology Quality of Life Index – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.5.1 | Summary of Summary of SCORing Atopic Dermatitis – Actual, Change, and Percent Change from Baseline | |
| 14.2.5.2 | Summary of Summary of SCORing Atopic Dermatitis – Actual, Change, and Percent Change from Baseline | |
| 14.2.6.1 | Summary of Visual Analog Scale of Pruritus – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.6.2 | Summary of Visual Analog Scale of Pruritus – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.7.1 | Summary of Body Surface Area – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.7.2 | Summary of Body Surface Area – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.8.1 | Summary of Trans epidemal Water Loss – Actual, Change, and Percent Change from Baseline | ITT |
| 14.2.8.2 | Summary of Trans epidemal Water Loss – Actual, Change, and Percent Change from Baseline | PP |
| 14.2.9.1 | Summary of Total DGLA Concentrations – Actual and Change from Baseline by IGA results | ITT |
| 14.2.9.2 | Summary of Free DGLA Concentrations – Actual and Change from Baseline by IGA results | ITT |
| | Safety Tables | |
| 14.3.1.1 | Overall Summary of Adverse Events | SAF |
| 14.3.1.2 | Summary of Treatment-Emergent Adverse Events | SAF |
| 14.3.1.3 | Summary of Related Treatment-Emergent Adverse Events | SAF |
| 14.3.1.4 | Summary of Treatment-Emergent Adverse Events by Severity | SAF |
| 14.3.1.5 | Summary of Treatment-Emergent Adverse Events by Relationship | SAF |
| 14.3.1.6 | Summary of Treatment-Emergent Adverse Events by Relationship and Severity | SAF |
| 14.3.1.7 | Summary of Treatment-Emergent Adverse Events leading to treatment discontinuation | SAF |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

| Table Number | Title | Population |
|---|---|---|
| 14.3.1.8 | Summary of Serious Treatment-Emergent Adverse Events | SAF |
| 14.3.1.9 | Summary of Related Serious Treatment-Emergent Adverse Events | SAF |
| 14.3.4.1.1 | Summary of Clinical Safety Laboratory Results – Serum Chemistry | SAF |
| 14.3.4.1.2 | Shift Table Clinical Laboratory – Serum Chemistry | SAF |
| 14.3.4.2.1 | Summary of Clinical Laboratory – Hematology | SAF |
| 14.3.4.2.2 | Shift Table Clinical Laboratory – Hematology | SAF |
| 14.3.4.3.1 | Summary of Clinical Laboratory – Urinalysis (Continuous) | SAF |
| 14.3.4.3.2 | Shift Table Clinical Laboratory – Urinalysis (Continuous) | SAF |
| 14.3.4.3.3 | Summary of Clinical Laboratory – Urinalysis (Categorical) | SAF |
| 14.3.5 | Summary of Vital Signs | SAF |

Table 14.1.1
Summary of Subject Enrollment and Disposition
(All Subjects)

| | | Treatemen | | |
|---|---|---|---|---|
| Parameter | Statistic | DS107G | Placebo | -<br>Total |
| Number of Subjects Screened | N | | | xx |
| Number of Subjects Screen Failed | N | | | xx |
| Number of Subjects Randomized | N | XX | xx | xx |
| Number of Subjects in Safety Population <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects in the Intent-to-Treat Population <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects in the Per Protocol Population <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>1</sup> Percentages are based on the number of randomized subjects.

Note(s): The Safety (SAF) population includes all randomized subjects who received at least one dose of the medication, according to treatment received.

The Intent-To-Treat (ITT) population includes all randomized subjects, according to the randomized treatment.

The Per Protocol (PP) population includes all subjects who received at least one dose of the medication and who had at least one post-baseline evaluation on the primary endpoint of IGA with no significant protocol deviations.

Program: t14 1 1.SAS, Generated on DDMMMYYY HH:MM

Table 14.1.2 Summary of Visits Completed

| Parameter | Statistic | Treatem | Treatement Group | |
|---|---|---|---|---|
| | | DS107G | Placebo | _<br>Total |
| Number of Subjects in Safety Population <sup>1</sup> | N | XX | XX | XX |
| Screening | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 8/ET | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Follow up/Week 10 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects in Intent-to-treat Population <sup>2</sup> | N | xx | xx | XX |
| Screening | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 8/ET | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Follow up/Week 10 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Subjects in Per Protocol Population <sup>3</sup> | N | xx | xx | xx |
| Screening | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 8/ET | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Follow up/Week 10 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>1</sup> Percentages are based on the number of subjects in the safety population.

Program: t14 1 2.SAS, Generated on DDMMMYYY HH:MM

<sup>2</sup> Percentages are based on the number of subjects in the intent-to-treat population.

<sup>3</sup> Percentages are based on the number of subjects in the per protocol population.

Table 14.1.3 Summary of Study Completion

| Parameter | | Treatement Group | | |
|---|---|---|---|---|
| | Statistic | DS107G | Placebo | —<br>Total |
| Number of Subjects in Safety Population | N | XX | XX | XX |
| Completed the study <sup>1</sup> | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>5</sup> | x.xxx | | |
| Primary Reason for Discontinuation <sup>4</sup> | | | | |
| Withdrawal by subject | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol violation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Lost to follow-up | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event or SAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>6</sup> | X.XXX | | |
| Number of days in study | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | XX, XX | xx, xx | XX, XX |

<sup>1</sup> Percentages are based on the number of subjects in the safety population.

Note(s): Number of days in the study is calculated as the difference between the date of the last visit (Follow up/Week 10) and the informed consent date plus 1.

Program: t14 1 3.SAS, Generated on DDMMMYYY HH:MM

<sup>2</sup> Percentages are based on the number of subjects in the intent-to-treat population.

<sup>3</sup> Percentages are based on the number of subjects in the per protocol population.

<sup>4</sup> Percentages are based on the number of subjects who discontinued within each population.

<sup>5</sup> p-value from Fisher Exact test

<sup>6</sup> p-value from a Pearson's Chi-Square test (using exact statement)

Table 14.1.3 Summary of Study Completion

| Parameters | Statistic | Treatement Group | | |
|---|---|---|---|---|
| | | DS107G | Placebo | <br>Total |
| Number of Subjects in Intent-to-treat Population | N | XX | XX | XX |
| Completed the $study^2$ | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>5</sup> | X.XXX | | |
| Primary Reason for Discontinuation <sup>4</sup> | | | | |
| Withdrawal by subject | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol violation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event or SAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | n (용) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (용) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>6</sup> | x.xxx | | |
| Number of days in study | n | XX | xx | XX |
| | Mean | XX.X | xx.x | XX.X |
| | SD | xx.x | XX.X | XX.X |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | xx, xx | xx, xx | XX, XX |

<sup>1</sup> Percentages are based on the number of subjects in the safety population.

Note(s): Number of days in the study is calculated as the difference between the date of the last visit (Follow up/Week 10) and the informed consent date plus 1.

Program: t14 1 3.SAS, Generated on DDMMMYYY HH:MM

<sup>2</sup> Percentages are based on the number of subjects in the intent-to-treat population.

<sup>3</sup> Percentages are based on the number of subjects in the per protocol population.

<sup>4</sup> Percentages are based on the number of subjects who discontinued within each population.

<sup>5</sup> p-value from Fisher Exact test

<sup>6</sup> p-value from a Pearson's Chi-Square test (using exact statement)

Table 14.1.3 Summary of Study Completion

| Parameters | Statistic | Treatement Group | | |
|---|---|---|---|---|
| | | DS107G | Placebo | —<br>Total |
| Number of Subjects in Per Protocol Population | N | XX | XX | XX |
| Completed the study <sup>3</sup> | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>5</sup> | x.xxx | , , | , |
| Primary Reason for Discontinuation <sup>4</sup> | | | | |
| Withdrawal by subject | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol violation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event or SAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>6</sup> | X.XXX | | |
| Number of days in study | n | xx | xx | xx |
| | Mean | XX.X | xx.x | XX.X |
| | SD | xx.x | xx.x | XX.X |
| | Median | xx.x | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | xx, xx | xx, xx | XX, XX |

<sup>1</sup> Percentages are based on the number of subjects in the safety population.

Note(s): Number of days in the study is calculated as the difference between the date of the last visit (Follow up/Week 10) and the informed consent date plus 1.

Program: t14 1 3.SAS, Generated on DDMMMYYY HH:MM

<sup>2</sup> Percentages are based on the number of subjects in the intent-to-treat population.

<sup>3</sup> Percentages are based on the number of subjects in the per protocol population.

<sup>4</sup> Percentages are based on the number of subjects who discontinued within each population.

<sup>5</sup> p-value from Fisher Exact test

<sup>6</sup> p-value from a Pearson's Chi-Square test (using exact statement)

Table 14.1.4
Summary of Protocol Deviations
(Safety Population)

| Deviations | | Treatement Group | | |
|---|---|---|---|---|
| | Statistic | DS107G<br>(N=XX) | Placebo<br>(N=XX) | Total (N=XX) |
| Missed dose(s) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Extra dose(s) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Fasting period not respected | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Randomization error | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study product not kept within temperature range | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study visit not done | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Visit performed out of window | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Procedure(s) done but not required by the protocol | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time window/order/of events for study procedure not respected | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study procedure(s) not done | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prohibithed Medications | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): n = Number of subjects. Each subject is counted only once within each deviation.

Program: t14\_1\_4.SAS, Generated on DDMMMYYY HH:MM
Table 14.1.5.1
Summary of Subject Demographics and Baseline Characteristics (Safety Population)

| | | Treateme | | |
|---|---|---|---|---|
| Characteristic | - | DS107G | Placebo | —<br>Total |
| | Statistic | (N=XX) | (N=XX) | (N=XX) |
| _ | (0) | , | , | , , |
| Sex | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | | | | |
| uge (years) | n | XX | xx | XX |
| | Mean | xx.x | xx.x | XX.X |
| | SD | xx.x | xx.x | XX.X |
| | Median | xx.x | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | XX, XX | XX, XX | xx, xx |
| Race | | | | |
| American Indian/Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Program: t14\_1\_5\_1.SAS, Generated on DDMMMYYY HH:MM

Table 14.1.5.1
Summary of Subject Demographics and Baseline Characteristics (Safety Population)

| | | Treateme | | |
|----------------|---------------|----------|---------|------------|
| | _ | DS107G | Placebo | -<br>Total |
| Characteristic | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Height (cm) | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | xx, xx | xx, xx | XX, XX |
| eight (kg) | n | xx | xx | XX |
| | Mean | xx.x | xx.x | XX.X |
| | SD | xx.x | xx.x | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Interquartile | xx, xx | xx, xx | xx, xx |
| MI (kg/m2) | n | xx | xx | XX |
| . 5 | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Interquartile | xx, xx | xx, xx | xx, xx |

Program: t14 1 5 1.SAS, Generated on DDMMMYYY HH:MM

| Table 14.1.5.2 | Summary | of | Subject | Demographics | and | Baseline | Characteristics | (Inte | ent-to-Tre | eat | Population |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Table 14.1.5.3 | Summary | of | Subject | Demographics | and | Baseline | Characteristics | (Per | Protocol | Pop | ulation) |

Table 14.1.6
Summary of Medical History
(Safety Population)

| Body System | | Treateme | | |
|-----------------------|-----------|-----------|-----------|------------|
| | | DS107G | Placebo | -<br>Total |
| | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Eyes-Ears-Nose-Throat | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Respiratory - Asthma | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Respiratory - Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cardiovascular | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gastrointestinal | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hepatobiliary | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Genitourinary/Renal | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reproductive | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neurological | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Endocrinal | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Hematological | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Musculoskeletal | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dermatological | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Extremities | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Immunological | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Psychiatric | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Allergies | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Program: t14\_1\_6.SAS, Generated on DDMMMYYY HH:MM

Table 14.1.7.1
Summary of Study Drug Exposure and Compliance (Safety Population)

| | | Treateme | | |
|------------------------|---------------|----------|------------|------------|
| | <del>-</del> | DS107G | Placebo | -<br>Total |
| Parameters | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Number of days on drug | | xx | ww | 22 |
| Number of days on drug | n<br>Mean | XX.X | XX<br>XX.X | XX<br>XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | xx, xx | xx, xx | xx, xx |
| Compliance (%) | n | xx | xx | xx |
| Compilance (%) | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | XX, XX | XX, XX | XX, XX |

Note(s): Number of days on drug is defined as (Date of Week 8/ET Visit - First dose of study drug administration date)

Compliance is defined as 100\*[(Sum of all capsules dispensed) - (Sum of all capsules returned)]/[4 x Number of days on drug]

Program: t14 1 7 1.SAS, Generated on DDMMMYYY HH:MM

| Table 14.1.7.2 | Summary | of | Study | Drug | Exposure | and | Compliance | (Intent-to-Treat Population) |
|---|---|---|---|---|---|---|---|---|
| Table 14.1.7.3 | Summary | οf | Study | Drua | Exposure | and | Compliance | (Per Protocol Population) |

Table 14.2.1.1.1

Summary of Investigator's Global Assessment - Responder Analysis at Week 8

(Intent-to-Treat Population)

| | | Treateme | | |
|---|---|---|---|---|
| | | DS107G | Placebo | <del>-</del><br>Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| IGA Score | | | | |
| Baseline | (0) | , | , | , |
| 3 - Moderate | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 - Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 - Very Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 8 | | | | |
| 0 - Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Almost Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Mild | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Moderate | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 - Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 - Very Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Responders <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | | | |
| Non-Responders | • • | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>2</sup> | X.XXX | | |
| | p-value <sup>3</sup> | x.xxx | | |
| Week 8 - Very Severe/Severe4 | | | | |
| 0 - Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Almost Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Mild | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Moderate | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 - Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 - Very Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Responders <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-Responders | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non Nospondors | p-value <sup>2</sup> | x. (xx.x)<br>x.xxx | ΔΑ (ΔΑ•Δ) | AA (AA•A) |
| AP version FINAL 1.0: DS107G-02 | 19 OCT 2015 | | P: | age 43 of 107 |

| Week 8 - Moderate <sup>4</sup> | | | | |
|--------------------------------|-------|-----------|-----------|-----------|
| 0 - Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Almost Clear | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Mild | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Moderate | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 - Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 - Very Severe | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Responders <sup>1</sup> | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-Responders | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

p-value<sup>2</sup>

x.xxx

Program: t14 2 1 1 1.SAS, Generated on DDMMMYYY HH:MM

<sup>1</sup> Subject is classified as Responder if he/she achieves an IGA score of 0 (clear) or 1 (almost clear) at Week 8

<sup>2</sup> p-value from a Cochran-Mantel-Haenszel test with site included as a stratification factor

<sup>3</sup> p-value from a Fisher Exact test (data from all sites combined)

<sup>4</sup> IGA score at baseline visit.

| Table 14.2.1.1.2 | Summary of Investigator's Global Assessment - Responder Analysis at Week 8 (Per Protocol Population) |
|---|---|
| Table 14.2.1.1.3 | Summary of Investigator's Global Assessment - Responder Analysis at Week 8 (Intent-to-Treat Population) Supportive Analysis (LOCF) |
| Table 14.2.1.1.4 | Summary of Investigator's Global Assessment - Responder Analysis at Week 8 (Per Protocol Population) Supportive Analysis (LOCF) |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Table 14.2.1.2.1

Summary of Investigator's Global Assessment - Actual, Change and Percent Change from Baseline (Intent-to-Treat Population)

Page 1 of 2

| | | Treateme | | |
|---|---|---|---|---|
| | | DS107G | Placebo | Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| IGA Score | | | | |
| Danalina | _ | | | |
| Baseline | n<br>Mean | XX | XX | XX |
| | SD | XX.X<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | xx, xx | xx, xx | xx, xx |
| Week 2 | 11124 | , | , | , |
| Actual | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | xx.x |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | xx, xx | xx, xx | xx, xx |
| Change from Baseline | n | XX | XX | xx |
| - | Mean | xx.x | xx.x | xx.x |
| | SD | XX.X | xx.x | XX.X |
| | Median | XX.X | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Interquartile | xx, xx | XX, XX | xx, xx |
| | ${	t LSMEANS^1}$ | XX.X | xx.x | |
| | 95% CI | (xx.x, xx.x) | (xx.x, xx.x) | |
| | p-value <sup>1</sup> | (,, | (, | |
| Percent Change from Baseline | n | xx | XX | XX |
| mange from baseline | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | | | |
| | Incerqualcite | xx, xx | xx, xx | XX, XX |

NOTE: Results at Week 4, Week 8, and Week 10 will also be presented as well as the change from Week 8 to Week 10.

1 LSMEANs and p-value from an ANCOVA on the change from baseline. The model includes Treatment group, Site as fixed effects and the baseline value as the covariate.

Note(s): Baseline is the result measured at Baseline Visit.

Program: t14 2 1 2 1.SAS, Generated on DDMMMYYY HH:MM

| Table 14.2.1.2.2 | Summary of Investigator's Global Assessment - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
|---|---|
| Table 14.2.2.1 | Summary of Eczema Area and Severity Index - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.2.2 | Summary of Eczema Area and Severity Index - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.3.1 | Summary of Patient-Oriented Eczema Measure - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.3.2 | Summary of Patient-Oriented Eczema Measure - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.4.1 | Summary of Dermatology Quality of Life Index - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.4.2 | Summary of Dermatology Quality of Life Index - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.5.1 | Summary of Summary of SCORing Atopic Dermatitis - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.5.2 | Summary of Summary of SCORing Atopic Dermatitis - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.6.1 | Summary of Visual Analog Scale of Pruritus - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.6.2 | Summary of Visual Analog Scale of Pruritus - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.7.1 | Summary of Body Surface Area - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.7.2 | Summary of Body Surface Area - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |
| Table 14.2.8.1 | Summary of Trans epidemal Water Loss - Actual, Change, and Percent Change from Baseline (Intent-to-Treat Population) |
| Table 14.2.8.2 | Summary of Trans epidemal Water Loss - Actual, Change, and Percent Change from Baseline (Per Protocol Population) |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Protocol No. DS107G-02

Table 14.2.1.3.1 Summary of Investigator's Global Assessment - Proportion of Subjects with at least 1-point decrease, and with no change or increase/decrease at Week 8 and Week 10 (Intent-to-Treat Population)

Page 1 of 1

| | | Treateme | | |
|---|---|---|---|---|
| | | DS107G | Placebo | _<br>Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| IGA Score | | | | |
| Week 8 | | | | |
| At least a 1-point decrease from baseline in IGA | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>1</sup> | x.xxx | | |
| Change from Baseline in IGA | | | | |
| 3-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No change | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| 2-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Week 10 | | | | |
| At least a 1-point decrease from baseline in IGA | | | | |
| Yes | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | p-value <sup>1</sup> | x.xxx | | |
| Change from Baseline in IGA | <del>-</del> | | | |
| 3-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-point decrease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No change | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| 2-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3-point increase | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>1</sup> p-value from a Cochran-Mantel-Haenszel test with site included as a stratification factor Note(s): Baseline is the result measured at Baseline Visit.

Program: t14 2 1 3 1.SAS, Generated on DDMMMYYY HH:MM

Table 14.2.1.3.2 Summary of Investigator's Global Assessment - Proportion of Subjects with at least 1-point decrease, and with no change or increase/decrease at Week 8 and Week 10 (Per Protocol Population)

Dignity Sciences


| | | | Treatement | Group | | | |
|---|---|---|---|---|---|---|---|
| | | DS10 | 7 G | Place | 00 | Tot | al |
| | | (N=XX | ₹) | (N=XX | ) | (N=> | XX) |
| Parameter | | | - | IGA Responde | r status¹ | | |
| Total DGLA | | Responder | Non<br>Responder | Responder | Non<br>Responder | Responder | Non<br>Responder |
| | Statistic | | | | | | |
| Baseline | n | | XX | | XX | | XX |
| | Mean | | XX.X | | XX.X | | XX.X |
| | SD | | XX.X | | XX.X | | XX.X |
| | Median | | XX.X | | XX.X | | XX.X |
| | Min, Max | | XX, XX | | XX, XX | | XX, XX |
| | Interquartile | | xx, xx | | xx, xx | | xx, xx |
| Week 4 | | | | | | | |
| Actual | n | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Median | XX.X | XX.X | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Interquartile | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Change from Baseline | n | xx | xx | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Interquartile | XX, XX | xx, xx | xx, xx | XX, XX | xx, xx | xx, xx |

NOTE: Results at Week 8 will also be presented as well as the change from Week 8 for DGLA result by IGA results at Week 10.

Note(s): Baseline is the nearest value to and before the first dose of the study medication.

Program: t14 2 9 1.SAS, Generated on DDMMMYYY HH:MM

<sup>&</sup>lt;sup>1</sup>IGA resuls for the corresponding visit

Table 14.2.9.2 Summary of Free DGLA Concentrations - Actual and Change from Baseline by IGA results (Intent-to-treat Population)

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Table 14.3.1.1

Overall Summary of Adverse Events (Safety Population)

| | | Treateme | | |
|---|---|---|---|---|
| Parameter | Statistic <sup>1</sup> | DS107G<br>(N=XX) | Placebo (N=XX) | Total (N=XX) |
| Number of Subjects with Treatment-Emergent Adverse Events | n(%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Number of Subjects with Related Treatment-Emergent Adverse Events | n(%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Number of Subjects with Serious Treatment-Emergent Adverse Events | n(%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Number of Subjects with Related Serious Treatment-Emergent Adverse Events | n(%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Number of Subjects with Treatment-Emergent Adverse Events leading to treatment discontinuation | n(%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

<sup>1</sup> n=number of subjects; E=number of events

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0)

Program: t14\_3\_1\_1.SAS, Generated on DDMMMYYY HH:MM

Table 14.3.1.2

Summary of Treatment-Emergent Adverse Events (Safety Population)

| | | Treateme | | |
|---|---|---|---|---|
| System Organ Class | <del>-</del> | DS107G | Placebo | Total<br>(N=XX) |
| Preferred Term | Statistic | (N=XX) | (N=XX) | |
| Number of subjects with at least one TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| OC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). Subjects experiencing the same adverse event multiple times within the same system organ class are counted only once for that system organ class. Similarly, subjects experiencing the same adverse event multiple times within the same preferred term are counted only once. Adverse events are sorted alphabetically by system organ class and within each system organ class, the preferred terms are presented by decreasing order of total frequency.

Program: t14 3 1 2.SAS, Generated on DDMMMYYY HH:MM

| Table 14.3.1.3 | Summary of Related Treatment-Emergent Adverse Events (Safety Population) |
|---|---|
| Table 14.3.1.7 | Summary of Treatment-Emergent Adverse Events leading to treatment discontinuation (Safety Populaiton |
| Table 14.3.1.8 | Summary of Serious Treatment-Emergent Adverse Events (Safety Population) |
| Table 14.3.1.9 | Summary of Related Serious Treatment-Emergent Adverse Events (Safety Population) |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Table 14.3.1.4

Summary of Treatment-Emergent Adverse Events by Severity (Safety Population)

| | | | | Treatement | Group | | |
|---|---|---|---|---|---|---|---|
| | | | DS107G | | | Placebo | |
| System Organ Class | | | (N=XX) | | | (N=XX) | |
| Preferred Term | Statistic | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Number of subjects with at least one TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). Subjects experiencing the same adverse event multiple times within the same system organ class are counted only once according to the highest severity for that system organ class. Similarly, subjects experiencing the same adverse event multiple times within the same preferred term are counted only once according to the highest severity. Adverse events are sorted alphabetically by system organ class and within each system organ class, the preferred terms are presented by decreasing order of total frequency.

Program: t14 3 1 4.SAS, Generated on DDMMMYYY HH:MM

Table 14.3.1.5

Summary of Treatment-Emergent Adverse Events by Relationship (Safety Population)

| | | Treatement Group | | | |
|---|---|---|---|---|---|
| | <del>-</del> | DS | 107G | Pla | acebo |
| Sustan Organ Class | _ | (N | =XX) | (N | =XX) |
| System Organ Class Preferred Term | Statistic | Related | Not Related | Related | Not Related |
| Number of subjects with at least one TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 50C2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). Subjects experiencing the same adverse event multiple times within the same system organ class are counted only once according to the greatest reported relationship for that system organ class. Similarly, subjects experiencing the same adverse event multiple times within the same preferred term are counted only once according to the greatest reported relationship. Adverse events are sorted alphabetically by system organ class and within each system organ class, the preferred terms are presented by decreasing order of total frequency.

Program: t14 3 1 5.SAS, Generated on DDMMMYYY HH:MM


 ${\small \mbox{Table 14.3.1.6}} \\ {\small \mbox{Summary of Treatment-Emergent Adverse Events by Relationship and Severity}} \\ ({\small \mbox{Safety Population}})$ 

| | | | | Treat | tement Group | | |
|---|---|---|---|---|---|---|---|
| | | | | | DS107G | | |
| | | | | | (N=XX) | | |
| | | M | ild | Mod | lerate | Se | vere |
| System Organ Class | | | | | | | |
| Preferred Term | Statistic | Related | Not Related | Related | Not Related | Related | Not Related |
| Number of subjects with at least one TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| OC2 | n (응) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). Subjects experiencing the same adverse event multiple times within the same system organ class are counted only once Term by using (1) the greatest reported relationship followed by (2) the highest reported intensity for that system organ class. Similarly, subjects experiencing the same adverse event multiple times within the same preferred term are counted only once Term by using (1) the greatest reported relationship followed by (2) the highest reported intensity. Adverse events are sorted alphabetically by system organ class and within each system organ class, the preferred terms are presented by decreasing order of total frequency.

Program: t14 3 1 6.SAS, Generated on DDMMMYYY HH:MM

 ${\small \mbox{Table 14.3.1.6}} \\ {\small \mbox{Summary of Treatment-Emergent Adverse Events by Relationship and Severity}} \\ ({\small \mbox{Safety Population}})$ 

| | | | | Treat | ement Group | | |
|---|---|---|---|---|---|---|---|
| | | | | | Placebo | | |
| | | | | | (N=XX) | | |
| | | М | ild | Mod | erate | Se | vere |
| System Organ Class | | | | | | | |
| Preferred Term | Statistic | Related | Not Related | Related | Not Related | Related | Not Related |
| Number of subjects with at least<br>one TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). Subjects experiencing the same adverse event multiple times within the same system organ class are counted only once Term by using (1) the greatest reported relationship followed by (2) the highest reported intensity for that system organ class. Similarly, subjects experiencing the same adverse event multiple times within the same preferred term are counted only once Term by using (1) the greatest reported relationship followed by (2) the highest reported intensity. Adverse events are sorted alphabetically by system organ class and within each system organ class, the preferred terms are presented by decreasing order of total frequency.

Program: t14 3 1 6.SAS, Generated on DDMMMYYY HH:MM

Table 14.3.4.1.1
Summary of Clinical Laboratory - Serum Chemistry (Safety Population)

| | | Treateme | nt Group | |
|---|---|---|---|---|
| | _ | DS107G | Placebo | -<br>Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| ALT (IU/L ) | | | | |
| Screening | n | xx | xx | XX |
| Actual | Mean | xx.x | xx.x | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | xx, xx | XX, XX |
| | Interquartile | XX, XX | xx, xx | XX, XX |
| Baseline | | | | |
| Actual | n | XX | XX | Xx |
| | Mean | XX.X | xx.x | XX.X |
| | SD | xx.x | xx.x | XX.X |
| | Median | xx.x | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| | Interquartile | xx, xx | xx, xx | XX, XX |
| Week 4 | | | | |
| Actual | n | XX | XX | XX |
| | Mean | xx.x | XX.X | XX.X |
| | SD | XX.X | xx.x | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| | Interquartile | xx, xx | XX, XX | XX, XX |
| Change from Baseline | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | |
| | Interquartile | xx, xx<br>xx, xx | xx, xx<br>xx, xx | XX, XX |

 $\underline{\text{NOTES}}$ : Results at Week 8 will also be presented. See Table  $\overline{1}$  for details on parameters to be presented

Note(s): Baseline is the nearest value to and before the first dose of the study medication.

Program: t14\_3\_4\_1\_1.SAS, Generated on DDMMMYYY HH:MM

Table 14.4.2.1 Summary of Clinical Laboratory - Hematology (Safety Population)

Table 14.4.3.1 Summary of Clinical Laboratory - Urinalysis (Continuous) (Safety Population)

Table 14.3.4.1.2
Shift Table Clinical Laboratory - Serum Chemistry (Safety Population)

| | | Treatement Group | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | DS107G | | | Placebo | |
| | Post-Baseline | Statistic | | (N=XX) | | | (N=XX) | |
| | Laboratory<br>Evaluation | | Baselin | e Laboratory Eva | aluation | Baseline | e Laboratory Ev | aluation |
| Parameter | | | Low | Normal | High | Low | Normal | High |
| ALT (IU/L ) | | | | | | | | |
| Week 4 | Low<br>Normal<br>High | n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Week 8 | Low<br>Normal<br>High | n (%)<br>n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

NOTE: See Table 1 for details on parameters to be presented.

Note(s): Baseline is the nearest value to and before the first dose of the study medication.

Program: t14\_3\_4\_1\_2.SAS, Generated on DDMMMYYY HH:MM

Table 14.4.2.2 Shift Table Clinical Laboratory - Hematology (Safety Population)

Table 14.4.3.2 Shift Table Clinical Laboratory - Urinalysis (Continuous) (Safety Population)


| | | Treateme | nt Group | |
|-----------|-----------|----------------|-----------|------------|
| | | DS107G Placebo | | —<br>Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Bilirubin | | | | |
| Screening | | | | |
| Positive | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Baseline | | | | |
| Positive | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Jeek 4 | | | | |
| Positive | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Jeek 8 | | | | |
| Positive | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Negative | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Program: t14\_3\_4\_3\_3.SAS, Generated on DDMMMYYY HH:MM

Table 14.3.5 Summary of Vital Signs (Safety Population)

| | | Treateme | nt Group | |
|---|---|---|---|---|
| | _ | DS107G | Placebo | -<br>Total |
| Parameter | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Systolic Blood Pressure (mmHg) | | | | |
| Screening | n | XX | xx | xx |
| Actual | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Interquartile | xx, xx | xx, xx | xx, xx |
| Baseline | | | | |
| Actual | n | XX | xx | Xx |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Interquartile | XX, XX | XX, XX | XX, XX |
| Week 2 | 1 | , | • | , |
| Actual | n | xx | xx | XX |
| | Mean | xx.x | xx.x | XX.X |
| | SD | xx.x | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | XX, XX | XX, XX |
| | Interquartile | xx, xx | xx, xx | XX, XX |
| Change from Baseline | n | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | | | |
| | | XX, XX | XX, XX | XX, XX |
| | Interquartile | XX, XX | XX, XX | XX, XX |

NOTES: Results at Week 4 and Week 8 will also be presented. All parameters (systolic/diastolic blood pressure, pulse, oral temperature and respiratory rate) all be presented.

Note(s): Baseline is the nearest value to and before the first dose of the study medication.

Program: t14\_3\_5.SAS, Generated on DDMMMYYY HH:MM

## 13.2 Mock Listings

The list of listings is presented in the table below followed by the actual mock listings. In all listings will appear the subject identification and the population indicator. They will be sorted by treatment group, study site, subject, and visit (when applicable).

| Listing | Title | Population |
|------------|-------------------------------------------|-----------------|
| Number | | |
| | Study Conduct Listings | |
| 16.2.1.1.1 | Subject Disposition | Screen Failures |
| 16.2.1.1.2 | Subject Disposition | Enrolled |
| 16.2.1.2 | Subject Visits | Enrolled |
| 16.2.2 | Protocol Deviations | Enrolled |
| 16.2.3 | Analysis Populations | Enrolled |
| 16.2.4.1 | Demographics and Baseline Characteristics | Enrolled |
| 16.2.4.2 | Medical History | Enrolled |
| 16.2.4.3 | Prior and Concomitant Medications | Enrolled |
| 16.2.4.4 | Other Procedures | Enrolled |
| 16.2.4.5 | Emollient | Enrolled |
| 16.2.5.1 | Study Drug Administration | Enrolled |
| 16.2.5.2 | Drug Accountability | Enrolled |
| 16.2.5.3 | Subject Compliance Log | Enrolled |
| 16.2.5.4 | Study Drug Exposure and Compliance | Enrolled |
| 16.2.5.5 | Total and Free DGLA plasma concentrations | Enrolled |
| | Efficacy Listings | |
| 16.2.6.1 | Investigator's Global Assessment | Enrolled |
| 16.2.6.2 | Eczema Area and Severity Index | Enrolled |
| 16.2.6.3 | Patient-Oriented Eczema Measure | Enrolled |
| 16.2.6.4 | Dermatology Quality of Life Index | Enrolled |
| 16.2.6.5 | SCORing Atopic Dermatitis | Enrolled |
| 16.2.6.6 | Trans epidemal Water Loss | Enrolled |
| | Safety Listings / Other Listings | |
| 16.2.7 | Adverse Events | Enrolled |
| 16.2.8.1 | Clinical Laboratory | Enrolled |
| 16.2.8.2 | Clinical Laboratory – Abnormal Results | Enrolled |
| 16.2.9 | Vital Signs | Enrolled |
| 16.2.10 | Physical Examination | Enrolled |
| 16.2.11 | Additional Information | Enrolled |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Lisintg 16.2.1.1.1 Subject Disposition (Screen Failed Subjects)

| | | | Meet All<br>Inclusion/Exclusion | |
|---|---|---|---|---|
| Site ID | Subject ID | Signature ICF | Criteria | Criteria Not Meet |

Program: L16\_2\_1\_1\_1.SAS, Generated on DDMMMYYY HH:MM

Lisintg 16.2.1.1.2 Subject Disposition (Enrolled Subjects)

| Treatment | | | Signature | Randomization | | Completed | Date of Completion/ | Primary Reason for |
|---|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | ICF | Date | Number | the study? | Discontinuation | Discontinuation |

Program: L16\_2\_1\_1\_2.SAS, Generated on DDMMMYYY HH:MM

Lisintg 16.2.1.2 Subject Visits (Enrolled Subjects)

| Treatment | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Screening | Baseline | Week 2 | Week 4 | Week 8/ET | Follow up/Week 10 |

Program: L16\_2\_1\_2.SAS, Generated on DDMMMYYY HH:MM

Lisintg 16.2.2 Protocol Deviations (Enrolled Subjects)

| Treatment | | | | | | | |
|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Date Reported ( | Category | Deviation | Impact |

Program: L16\_2\_2.SAS, Generated on DDMMMYYY HH:MM

Lisintg 16.2.3 Analysis Population (Enrolled Subjects)

| | | | | | | Reason not included in |
|---|---|---|---|---|---|---|
| | | | Intent-to- | | | Intent-to-treat Population/ |
| Treatment | | | Treat | Safety | Per Protocol | Safety Population/ |
| Group | Site ID | Subject ID | Population | Populaiton | Population | Per Protocol Population |

Program: L16\_2\_3.SAS, Generated on DDMMMYYY HH:MM

Lisintg 16.2.4.1
Demographic and Baseline Characteristics
(Enrolled Subjects)

| Treatment | Site ID | | | | | | Ethnicity | Height (cm) | Weight (kg) | BMI (kg/m2) |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | DICC ID | Subject ID | DOB | Age (years) | Gender | Race | псиитетей | neigne (em) | Weight (kg) | Dit (Rg/IIIZ) |

Program: L16\_2\_4\_1.SAS, Generated on DDMMMYYY HH:MM
Dignity Sciences

Lisintg 16.2.4.2 Medical History (Enrolled Subjects)

| | | | | | | | | Improved | Improved |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | from | from |
| | | | | | | | | Baseline at | Baseline at |
| Treatment | | | | | Onset | | Resolution | Week 8 | Week 10 |
| Group | Site ID | Subject ID | Body System | Medical/Surgical term | Date | Ongoing | Date | Visit | Visit |

Lisintg 16.2.4.3
Prior and Concomitant Medications
(Enrolled Subjects)

| | | | | | Dose/ | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | | | Medication/ | | Freq/ | | | | Prior or |
| Group | Site ID | Subject ID | ATC Classification | Indication | Route | Start Date | Ongoing | Stop Date | Concomitant |

Note(s): Medications are coded using WHO-Drug dictionary (version June 2013 B2).

Lisintg 16.2.4.4 Other Procedures (Enrolled Subjects)

| Treatment | | | | | | | | Prior or |
|---|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Procedure | Indication | Start Date | Ongoing | Stop Date | Concomitant |

Lisintg 16.2.4.5 Emollient (Enrolled Subjects)

| - | | | | | | | |
|---|---|---|---|---|---|---|---|
| Treatment | | | | | | | Prior or |
| Group | Site ID | Subject ID | Emollient Name | Start Date | Ongoing | Stop Date | Concomitant |

Lisintg 16.2.5.1
Study Drug Admnistration
(Enrolled Subjects)

| Treatment | | | | Was Study Drug | | Administration | Administration |
|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Administered? | If no, Reason | Date | Time |

Lisintg 16.2.5.2 Drug Accountability (Enrolled Subjects)

| Treatment | | | | Date | | Capsules | Date | Capsules | |
|---|---|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Dispensed | Batch Number | Dispensed | returned | Returned | Comments |

Lisintg 16.2.5.3 Subject Compliance Log (Enrolled Subjects)

| | | | | Missing doses | If Yes, | |
|---|---|---|---|---|---|---|
| Treatment | | | | since last | Number of | |
| Group | Site ID | Subject ID | Visit | visit? | missed doses | Comment |

# Lisintg 16.2.5.4 Study Drug Exposure and Compliance (Enrolled Subjects)

| Treatment | | | Number of | |
|-----------|---------|------------|--------------|----------------|
| Group | Site ID | Subject ID | days on drug | Compliance (%) |

# Lisintg 16.2.5.5 Total and Free DGLA plasma concentrations (Enrolled Subjects)

| Treatment | | | | | |
|-----------|---------|------------|---------|-------|--------|
| Group | Site ID | Subject ID | Analyte | Visit | Result |

Lisintg 16.2.6.1
Investigator's Global Assessment
(Enrolled Subjects)

| Treatment | | | | |
|------------|---------|------------|-------|------------|
| TTEACHETIC | | | | |
| C | Site ID | Subject ID | Visit | Assessment |
| Group | | | | |

Dignity Sciences

Lisintg 16.2.6.2 (Part 1)
Eczema Area and Severity Index
(Enrolled Subjects)

| Treatment<br>Group | Site ID | Subject ID | Visit | Head | Upper<br>Extremities | Trunk | Lower<br>Extremities |
|---|---|---|---|---|---|---|---|

Dignity Sciences

Lisintg 16.2.6.2 (Part 2)
Eczema Area and Severity Index
(Enrolled Subjects)

| | | | | | Induration | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Site ID | Subject ID | Visit | Head | Upper<br>Extremities | Trunk | Lower<br>Extremities |

Lisintg 16.2.6.2 (Part 3)
Eczema Area and Severity Index
(Enrolled Subjects)

| | | | Excoria | ation | | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Site ID | Subject ID | Visit | Head | Upper<br>Extremities | Trunk | Lower<br>Extremities |

Dignity Sciences

Lisintg 16.2.6.2 (Part 4)
Eczema Area and Severity Index
(Enrolled Subjects)

| | | | | | Lichenification | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Site ID | Subject ID | Visit | Head | Upper<br>Extremities | Trunk | Lower<br>Extremities | EASI Score |

Dignity Sciences

Lisintg 16.2.6.3
Patient-Oriented Eczema Measure
(Enrolled Subjects)

| Treatment | a' | 0.1.1 | | Q1 | 0.0 | 22 | 0.4 | 0.5 | 0.6 | 0.7 | 20214 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | QI | Q2 | Q3 | Q4 | Q5 | Q6 | Q / | POEM Score |

Dignity Sciences

Lisintg 16.2.6.4 (Part 1)
Dermatology Quality of Life Index
(Enrolled Subjects)

| Treatment | a1 | 0.1.1 | | 0.1 | 0.0 | 2.2 | 0.4 | 0.5 | 0.6 |
|-----------|---------|------------|-------|-----|-----|-----|-----|-----|-----|
| Group | Site ID | Subject ID | Visit | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 |

Dignity Sciences

Lisintg 16.2.6.4 (Part 2)
Dermatology Quality of Life Index
(Enrolled Subjects)

| Treatment | Site ID | Subject ID | Wieit | 07 | 074 | 08 | 09 | 010 | DLQI Score |
|---|---|---|---|---|---|---|---|---|---|
| Group | DICC ID | bubjece ib | VISIC | 2 / | 2/11 | QU | 20 | 210 | DIQI DCOIC |

Dignity Sciences

Lisintg 16.2.6.5 (Part 1) SCORing Atopic Dermatitis (Enrolled Subjects)

| | | | | Ervthema | Edema/Papulation | Ooging/Crust | Evannintion | Tichonification | Dryness | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | | | | | | - | | | _ | |
| Group | Site ID | Subject ID | Visit | Intensity | Intensity | Intensity | Intensity | Intensity | Intensity | Intensity |

Dignity Sciences

Lisintg 16.2.6.5 (Part 2) SCORing Atopic Dermatitis (Enrolled Subjects)

| | | | | | | Sleep loss | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | | | | Extent | Pruritus VAS | VAS Symptom | Objective | |
| Group | Site ID | Subject ID | Visit | Area involved (BSA) | Symptom Score | Score | SCORAD | SCORAD |

# Lisintg 16.2.6.6 Trans Epithelial Water Loss (Enrolled Subjects)

| | | | | | | | | Control |
|---|---|---|---|---|---|---|---|---|
| Treatment | | | | | | Measurement | | Measurement |
| Group | Site ID | Subject ID | Visit | Area | Represented Area | (g/m2h) | Control Area | (g/m2h) |

Lisintg 16.2.7 Adverse Events (Enrolled Subjects)

| | | System Organ Class/ | | | | | Severity/ | Action | Action | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | | Preferred Term/ | | End | Onset | | Relationship/ | Taken | Taken | |
| Group | Subject ID | Verbatim | Onset Date | Date | Day | Dur. | Outcome | Drug | Subject | SAE |

Note(s): Adverse events are coded using MedDRA dictionary (version 17.0). \*Treatment-Emergent Adverse Event. Dur.=Duration. Severity: Mild; Mod.= Moderate; Sev.=Severe. Relationship: Rel.=Related; Not Rel.=Not Related. Outcome: Rec/Res= Recovered/Resolved; Rec/Res. Seq= Recovered/Resolved with Sequelae; Recing/Resing= Recovering/Resolving; NotRec/NotRes= Not Recovered/ NotResolved; Unk=Unknown. Action Taken Drug: NotChg=Dose not changed; Inter.=Treatment interrupted; Withdr.=Treatment Withdrawn; NA=Not applicable; Unk.=Unknown; Oth.=Other. Action Taken Subject: NotReq=Not required; TrtUsed.=Treatment used; Withdr.=Subject Withdrawn; Unk.=Unknown; Oth.=Other.

Dignity Sciences

Lisintg 16.2.8.1 Clinical Laboratory (Enrolled Subjects)

| Treatment | | | | | Laboratory ' | Test | |
|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Category | (units) | Normal Range | Result |

Note(s): (L)=Below normal range; (H)=Above normal range

Dignity Sciences

Lisintg 16.2.8.2
Clinical Laboratory - Abnormal Results
(Enrolled Subjects)

| Treatment | | | | | Laboratory T | est | |
|---|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Category | (units) | Normal Range | Result |

Note(s): (L)=Below normal range; (H)=Above normal range

Dignity Sciences

Lisintg 16.2.9 Vital Signs (Enrolled Subjects)

| Treatment | | | | Parameter | |
|-----------|---------|------------|-------|-----------|--------|
| Group | Site ID | Subject ID | Visit | (units) | Result |

Lisintg 16.2.10
Physical Examination
(Enrolled Subjects)

| Treatment | | | | | | Description of |
|---|---|---|---|---|---|---|
| Group | Site ID | Subject ID | Visit | Body System | Results | Abnormality |

Lisintg 16.2.10
Physical Examination
(Enrolled Subjects)

| | | | Was there any | | | |
|---|---|---|---|---|---|---|
| Treatment | | | additional | | | |
| Group | Site ID | Subject ID | information | Visit | Form | Comments/Clarifications |

## 13.3 Mock Figures

The list of Figures is presented in the table below followed by the actual mock.

| Figure<br>Number | Title | Population |
|---|---|---|
| 14.2.1.1.1 | Bar Chart of the Number of Subjects on the Change from Baseline in IGA during study | ITT |
| 14.2.1.1.2 | Bar Chart of the Number of Subjects on the Change from Baseline in IGA during study | PP |
| 14.2.1.2.1 | Mean Change from baseline in IGA during study | ITT |
| 14.2.1.2.2 | Mean Change from baseline in IGA during study | PP |
| 14.2.1.3.1 | Mean Percent Change from baseline in IGA during study | ITT |
| 14.2.1.3.2 | Mean Percent Change from baseline in IGA during study | PP |
| 14.2.2.1.1 | Mean Change from baseline in EASI during study | ITT |
| 14.2.2.1.2 | Mean Change from baseline in EASI during study | PP |
| 14.2.2.2.1 | Mean Percent Change from baseline in EASI during study | ITT |
| 14.2.2.2.2 | Mean Percent Change from baseline in EASI during study | PP |
| 14.2.3.1.1 | Mean Change from baseline in POEM during study | ITT |
| 14.2.3.1.2 | Mean Change from baseline in POEM during study | PP |
| 14.2.3.2.1 | Mean Percent Change from baseline in POEM during study | ITT |
| 14.2.3.2.2 | Mean Percent Change from baseline in POEM during study | PP |
| 14.2.4.1.1 | Mean Change from baseline in DLQI during study | ITT |
| 14.2.4.1.2 | Mean Change from baseline in DLQI during study | PP |
| 14.2.4.2.1 | Mean Percent Change from baseline in DLQI during study | ITT |
| 14.2.4.2.2 | Mean Percent Change from baseline in DLQI during study | PP |
| 14.2.5.1.1 | Mean Change from baseline in SCORAD during study | ITT |
| 14.2.5.1.2 | Mean Change from baseline in SCORAD during study | PP |
| 14.2.5.2.1 | Mean Percent Change from baseline in SCORAD during study | ITT |
| 14.2.5.2.2 | Mean Percent Change from baseline in SCORAD during study | PP |
| 14.2.6.1.1 | Mean Change from baseline in VAS during study | ITT |
| 14.2.6.1.2 | Mean Change from baseline in VAS during study | PP |
| 14.2.6.2.1 | Mean Percent Change from baseline in VAS during study | ITT |
| 14.2.6.2.2 | Mean Percent Change from baseline in VAS during study | PP |
| 14.2.7.1.1 | Mean Change from baseline in BSA during study | ITT |
| 14.2.7.1.2 | Mean Change from baseline in BSA during study | PP |
| 14.2.7.2.1 | Mean Percent Change from baseline in BSA during study | ITT |
| 14.2.7.2.2 | Mean Percent Change from baseline in BSA during study | PP |

| nange from baseline in TEWL during study nange from baseline in TEWL during study ercent Change from baseline in TEWL during study | ITT<br>PP<br>ITT |
|---|---|
| nange from baseline in TEWL during study<br>ercent Change from baseline in TEWL during study | PP<br>ITT |
| ercent Change from baseline in TEWL during study | İTT |
| and Object of feet beautiful in TEVAL decision at adv | |
| ercent Change from baseline in TEWL during study | PP |
| Plot of Total DGLA concentrations at Baseline versus IGA score at Week 8 | ITT |
| Plot of Free DGLA concentrations at Baseline versus IGA score at Week 8 | ITT |
| Plot of Change from Baseline Total DGLA concentrations at Week 8versus IGA score at Week 8 | ITT |
| Plot of Change from Baseine Free DGLA concentrations at Week 8 versus IGA score at Week 8 | ITT |
| | ITT |
| · | ITT |
| | Plot of Free DGLA concentrations at Baseline versus IGA score at Week 8 Plot of Change from Baseline Total DGLA concentrations at Week 8 versus IGA score at Week 8 Plot of Change from Baseline Free DGLA concentrations at Week 8 versus IGA score at Week 8 Plot of Change from Baseline Total DGLA concentrations at Week 8 versus IGA score at Week 10 Plot of Change from Baseline Free DGLA concentrations at Week 8 versus IGA score at Week 10 |

Figure 14.2.1.1.1 Bar Chart of the Number of Subjects on the Change from Baseline in IGA during study (Intent-to-Treat Population)



Program: F14 2 1 1 1.SAS, Generated on DDMMMYYY HH:MM

#### Similar Figure will be provided for

14.2.1.1.2 Bar Chart of the Number of Subjects on the Change from Baseline in IGA during study (Per Protocol Population)

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 


Figure 14.2.1.2.1
Mean Change from baseline in IGA during study
(Intent-to-Treat Population)



Test ••• Reference

### Similar Figures will be provided for

| 14.2.1.2.2 | Mean Change from baseline in IGA during study (Per Protocol Population) |
|---|---|
| 14.2.1.3.1 | Mean Percent Change from baseline in IGA during study (Intent-to-Treat Population) |
| 14.2.1.3.2 | Mean Percent Change from baseline in IGA during study (Per Protocol Population) |
| 14.2.2.1.1 | Mean Change from baseline in EASI during study (Intent-to-Treat Population) |
| 14.2.2.1.2 | Mean Change from baseline in EASI during study (Per Protocol Population) |
| 14.2.2.2.1 | Mean Percent Change from baseline in EASI during study (Intent-to-Treat Population) |
| 14.2.2.2.2 | Mean Percent Change from baseline in EASI during study (Per Protocol Population) |
| 14.2.3.1.1 | Mean Change from baseline in POEM during study (Intent-to-Treat Population) |
| 14.2.3.1.2 | Mean Change from baseline in POEM during study (Per Protocol Population) |
| 14.2.3.2.1 | Mean Percent Change from baseline in POEM during study (Intent-to-Treat Population) |
| 14.2.3.2.2 | Mean Percent Change from baseline in POEM during study (Per Protocol Population) |
| 14.2.4.1.1 | Mean Change from baseline in DLQI during study (Intent-to-Treat Population) |
| 14.2.4.1.2 | Mean Change from baseline in DLQI during study (Per Protocol Population) |
| 14.2.4.2.1 | Mean Percent Change from baseline in DLQI during study (Intent-to-Treat Population) |
| 14.2.4.2.2 | Mean Percent Change from baseline in DLQI during study (Per Protocol Population) |
| 14.2.5.1.1 | Mean Change from baseline in SCORAD during study (Intent-to-Treat Population) |
| 14.2.5.1.2 | Mean Change from baseline in SCORAD during study (Per Protocol Population) |
| 14.2.5.2.1 | Mean Percent Change from baseline in SCORAD during study (Intent-to-Treat Population) |
| 14.2.5.2.2 | Mean Percent Change from baseline in SCORAD during study (Per Protocol Population) |
| 14.2.6.1.1 | Mean Change from baseline in VAS during study (Intent-to-Treat Population) |
| 14.2.6.1.2 | Mean Change from baseline in VAS during study (Per Protocol Population) |

| 14.2.6.2.1 | Mean Percent Change from baseline in VAS during study (Intent-to-Treat Population) |
|---|---|
| 14.2.6.2.2 | Mean Percent Change from baseline in VAS during study (Per Protocol Population) |
| 14.2.7.1.1 | Mean Change from baseline in BSA during study (Intent-to-Treat Population) |
| 14.2.7.1.2 | Mean Change from baseline in BSA during study (Per Protocol Population) |
| 14.2.7.2.1 | Mean Percent Change from baseline in BSA during study (Intent-to-Treat Population) |
| 14.2.7.2.2 | Mean Percent Change from baseline in BSA during study (Per Protocol Population) |
| 14.2.8.1.1 | Mean Change from baseline in TEWL during study (Intent-to-Treat Population) |
| 14.2.8.1.2 | Mean Change from baseline in TEWL during study (Per Protocol Population) |
| 14.2.8.2.1 | Mean Percent Change from baseline in TEWL during study (Intent-to-Treat Population) |
| 14 2 8 2 2 | Mean Percent Change from baseline in TEWI during study (Per Protocol Population) |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 

Figure 14.2.9.1
Scatter Plot of Total DGLA concentrations at Baseline versus IGA score at Week 8
(Intent-to-Treat Population)



Total DGLA Concentrations (Baseline)

### Similar Figures will be provided for

| 14.2.9.2 | Scatter Plot of Free DGLA concentrations at Baseline versus IGA score at Week 8 (Intent-to-Treat Population) |
|---|---|
| 14.2.10.1 | Scatter Plot of Change from Baseline Total DGLA concentrations at Week 8versus IGA score at Week 8 (Intent-to-Treat Population) |
| 14.2.10.2 | Scatter Plot of Change from Baseine Free DGLA concentrations at Week 8 versus IGA score at Week 8 (Intent-to-Treat Population) |
| 14.2.11.1 | Scatter Plot of Change fdrom Baseline Total DGLA concentrations at Week 8 versus IGA score at Week 10 (Intent-to-Treat Population |
| 14.2.11.2 | Scatter Plot of Change fdrom Baseline Free DGLA concentrations at Week 8 versus IGA score at Week 10 (Intent-to-Treat Population) |

SAP version FINAL 1.0: DS107G-02 19 OCT 2015 